CLINICAL TRIAL: NCT06943027
Title: Investigation of the Relationship Between Dysfunctional Breathing and Physical Fitness Parameters in Healthy Adults
Brief Title: Investigation of the Relationship Between Dysfunctional Breathing and Physical Fitness Parameters in Healty Adults
Acronym: DISFIT
Status: Not yet recruiting | Type: Observational
Sponsor: Elif Tunç (Other)
Responsible Party: Sponsor-Investigator, Elif Tunç, MS.c. PT, Istinye University
Organization: Istinye University (Other)
Other Study IDs: ISTU-DS-2025-ET; 2209-A (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey (TUBITAK))
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Dysfunctional Breathing
Keywords: ALPHA-FIT; Physical Fitness; Respiratory Function; MIP; MEP; Hyperventilation; Young Adults
MeSH Terms: conditions — Respiratory Aspiration; Hyperventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to investigate the relationship between dysfunctional breathing and physical fitness parameters in healthy adults aged 18-35. Participants will be evaluated using the Nijmegen Questionnaire to assess dysfunctional breathing symptoms, and their physical fitness will be measured using the ALPHA-FIT Test Battery. Respiratory muscle strength and pulmonary function will also be assessed. The findings may help healthcare professionals better understand dysfunctional breathing and develop targeted treatment programs.

DETAILED DESCRIPTION:
Dysfunctional breathing (DB) is characterized by chronic alterations in the respiratory cycle, often leading to symptoms such as dyspnea, chest tightness, and hyperventilation. Despite its prevalence, DB is frequently underdiagnosed and mismanaged due to limited awareness among healthcare professionals. This cross-sectional study aims to evaluate the relationship between DB symptoms and physical fitness in healthy young adults. A total of 38 participants diagnosed with DB will be assessed at Istinye University using the Nijmegen Questionnaire, ALPHA-FIT Test Battery, spirometry, and measurements of maximum inspiratory (MIP) and expiratory (MEP) mouth pressures. Data on sociodemographic characteristics will also be collected. The results of this study are expected to support clinicians in the accurate identification of DB and provide insight for the development of personalized rehabilitation strategies that improve physical fitness and respiratory health.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years
* Healthy individuals with no known systemic, neurological, or musculoskeletal disorders
* Nijmegen Questionnaire score >23 (indicative of dysfunctional breathing)
* Voluntary participation with informed consent

Exclusion Criteria:

* Diagnosed with respiratory, cardiovascular, or metabolic disease
* Currently receiving physiotherapy or pulmonary rehabilitation
* Regular use of medication affecting breathing or exercise capacity
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of healthy adults aged 18-35 years with no known systemic, neurological, or musculoskeletal conditions. Participants will be screened using the Nijmegen Questionnaire to identify symptoms of dysfunctional breathing.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Nijmegen Questionnaire Score | Baseline
  Assessment of dysfunctional breathing symptoms using the Nijmegen Questionnaire.

SECONDARY OUTCOMES:
ALPHA-FIT Test Battery Performance | Baseline
  Evaluation of physical fitness components such as strength, flexibility, balance, and endurance in participants.
Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP) | Baseline
  Measurement of respiratory muscle strength using a mouth pressure device to evaluate inspiratory and expiratory capacities.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kiesel K, Plisky PJ, Voight ML. Can Serious Injury in Professional Football be Predicted by a Preseason Functional Movement Screen? N Am J Sports Phys Ther. 2007 Aug;2(3):147-58. PMID 21522210
- [Background] Courtney R. The functions of breathing and its dysfunctions and their relationship to breathing therapy. Int J Osteopath Med. 2009;12(3):78-85. doi:10.1016/j.ijosm.2009.04.002
- See also: Review article on dysfunctional breathing and its assessment in physiotherapy. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4783243/